CLINICAL TRIAL: NCT04239573
Title: Comparing the Clinical Impact of Pancreatic Cyst Surveillance Programs
Brief Title: Comparing Two Methods to Follow Patients With Pancreatic Cysts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA2185; NCI-2019-04790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2185 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EA2185 (Other: DCP); EA2185 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (low intensity surveillance) (Experimental): Patients undergo MRI or CT at the beginning of the trial and again in 1 year. Following the first year, patients with no abnormalities repeat MRI or CT every 2 years. Patients with positive imaging features on MRI and CT at 1 or 2 years and with negative EUS, repeat MRI or CT in 1 year. Patients with negative imaging repeat MRI or CT in 2 years.
  Interventions: Procedure: Computed Tomography; Procedure: Endoscopic Ultrasound; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (high intensity surveillance) (Experimental): Patients undergo MRI or CT. Patients with 1-2 cm cyst undergo MRI or CT every 6 months for 1 year, then every 12 months for 2 years, and then every 24 months thereafter. Patients with 2-3 cm cyst undergo EUS within 6 months, and if EUS is negative, patients repeat MRI or CT in 1 year. If second EUS is negative, patients undergo alternate MRI or CT and EUS every 12 months. Patients with cyst > 3 cm undergo EUS within 6 months, and if EUS is negative, patients undergo alternate MRI or CT with EUS every 3-6 months.
  Interventions: Procedure: Computed Tomography; Procedure: Endoscopic Ultrasound; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT scan; Computerized Axial Tomography; computerized tomography; CT; CT scan; tomography
Procedure: Endoscopic Ultrasound — Undergo EUS
  Other Names: endosonography; EUS
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The purpose of this study is to compare the two approaches for monitoring pancreatic cysts. The study doctors want to compare more frequent monitoring vs less frequent monitoring in order to learn which monitoring method leads to better outcome for patients with pancreatic cysts.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of unfavorable clinical outcomes in the two arms.

SECONDARY OBJECTIVES:

I. To compare rates of major surgical morbidity and/or mortality between arms. II. To compare pancreatic cancer incidence and all-cause mortality across arms. III. Compare institutional (direct) costs. IV. Compare healthcare utilization of imaging, invasive testing, surgical, and other procedures across the two surveillance arms.

V. Compare patient (out-of-pocket and other indirect) costs. VI. Describe diagnostic test and treatment pathways by arm. VII. Compare patient reports of quality of life (QOL), situational anxiety. VIII. Compare patient report of financial distress. IX. Compare rates of non-adherence by arm assignment. X. To evaluate and compare the predictive performance of known and future biomarkers for dysplasia or cancer.

EXPLORATORY OBJECTIVE:

I. To evaluate and compare the predictive accuracy of known and future radiomic markers for dysplasia and pancreatic cancer.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (LOW INTENSITY SURVEILLANCE): Patients undergo magnetic resonance imaging (MRI) or computed tomography (CT) at the beginning of the trial and again in 1 year. Following the first year, patients with no abnormalities repeat MRI or CT every 2 years. Patients with positive imaging features on MRI and CT at 1 or 2 years and with negative endoscopic ultrasound (EUS), repeat MRI or CT in 1 year. Patients with negative imaging repeat MRI or CT in 2 years.

ARM B (HIGH INTENSITY SURVEILLANCE): Patients undergo MRI or CT. Patients with 1-2 cm cyst undergo MRI or CT every 6 months for 1 year, then every 12 months for 2 years, and then every 24 months thereafter. Patients with 2-3 cm cyst undergo EUS within 6 months, and if EUS is negative, patients repeat MRI or CT in 1 year. If second EUS is negative, patients undergo alternate MRI or CT and EUS every 12 months. Patients with cyst > 3 cm undergo EUS within 6 months, and if EUS is negative, patients undergo alternate MRI or CT with EUS every 3-6 months.

After completion of imaging procedures, patients are followed up for 5 years from the date of registration .

ELIGIBILITY:
* Patient must be ≥ 50 years and ≤ 75 years of age.
* Patient must not have acute pancreatitis or a history of chronic pancreatitis.
* Patient must have received a CT, MRI, or EUS within 6 months prior to randomization that revealed one or more ≥ 1 cm pancreatic cyst (s).
* Patients of childbearing potential must not be known to be pregnant.
* Patient must not have a prior diagnosis of pancreatic malignancy of any type.
* Patient must not have a history of pancreatic resection.
* Patients with only pancreatic lesions without malignant risk (pancreatic pseudocyst or classic serous cystic lesion) are not eligible.
* Patient must not have a family history of pancreatic adenocarcinoma in one or more first degree relatives(biological parents, full siblings or children).
* Patient must not have pancreatic cyst morphology that would prompt immediate surgical consideration (enhancing mural nodule, solid component in cyst, pancreatic duct ≥10mm, cyst causing obstructive jaundice).
* Patient must not have a comorbid illness that precludes pancreatic cyst resection.
* Patient must not be participating in any form of pancreatic cyst surveillance.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4606 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2037-06-03 (Estimated); Study Completion 2037-06-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an "unfavorable" outcome | Up to 5 years
  Defined as a composite of: (1) any pancreatic cancer without surgery; (2) unresectable pancreatic cancer or cancer > T1a, N0 at surgery, and (3) benign disease at surgery will be approached from the intent-to-treat perspective. Time to the first occurrence of the primary endpoint will measured from randomization. Survival analysis methods will be used to estimate and compare distributions of time to an unfavorable event between the study arms. In particular Kaplan-Meier estimates will be developed for each arm and a log rank test will be used to compare the two arms.

SECONDARY OUTCOMES:
Surgical and all-cause mortality | Up to 5 years
  Rates of major surgical morbidity and/or mortality will be estimated and compared across arms. All-cause mortality will be estimated and compared between the arms using log rank tests.
Major surgical morbidity | Up to 5 years
  Rates of major surgical morbidity and/or mortality will be estimated and compared across arms.
Pancreatic cancer incidence | Up to 5 years
  Pancreatic-cancer incidence and pancreatic cancer specific mortality will be estimated and compared between the arms using log rank tests.
Healthcare utilization of imaging, invasive testing, surgical, and other procedures using information collected from sites. | Up to 5 years
  Will compare between two arms.
Patient (out-of-pocket and other indirect) costs collected from patient surveys | Up to 5 years
  Will compare between two arms.
Patient reports of quality of life | Up to 5 years
  Will be assessed by Patient Reported Outcomes Measurement Information System10. Will compare between arms. Longitudinal regression modelling will be completed to account for the repeated assessments over time.
Patient reports of situational anxiety | Up to 5 years
  Will be assessed by Patient Reported Outcomes Measurement Information System-Anxiety short form. Will compare between arms.
Patient report of financial distress collected through patient surveys | Up to 5 years
  Will compare between arms.
Rates of non-adherence | Up to 5 years
  Will compare rates of non-adherence by arm assignment.
Biomarker analysis from collected samples to compare the predictive performance of known and future biomarkers for dysplasia or cancer | Up to 5 years
  Will evaluate and compare the predictive performance of known and future biomarkers for dysplasia or cancer.

OTHER OUTCOMES:
Predictive accuracy of radiomic markers for dysplasia and pancreatic cancer | Up to 5 years
  Will evaluate and compare the predictive accuracy of known and future radiomic markers for dysplasia and pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: David S Weinberg, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (352):
- United States (337):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Enloe Medical Center, Chico, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital-Hamden Care Center, Hamden, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale-New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Bromenn Lifecare Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - CentraState Medical Center, Freehold, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital - Monroe Campus, Stroudsburg, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Baptist Hospital, Columbia, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Alexandria Hospital, Alexandria, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Valley Health / Winchester Medical Center, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (4):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
- Puerto Rico (9):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan
- South Korea (2):
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Yonsei University Health System-Severance Hospital, Seoul

REFERENCES:
- [Derived] Weinberg DS, Gatsonis C, Zeh HJ, Carlos RC, O'Dwyer PJ; EA2185 Team. Comparing the clinical impact of pancreatic cyst surveillance programs: A trial of the ECOG-ACRIN cancer research group (EA2185). Contemp Clin Trials. 2020 Oct;97:106144. doi: 10.1016/j.cct.2020.106144. Epub 2020 Sep 10. PMID 32920242